CLINICAL TRIAL: NCT01366378
Title: A Phase 1, Open-Label, Study of the Effect of Cimetidine, a Known Inhibitor of Active Renal Secretion, on the Single-Dose Pharmacokinetics of Intravenously-Administered Methylnaltrexone in Healthy Adults
Brief Title: Effect of Cimetidine on the Single-Dose PK of IV- Administered MNTX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1304
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): methylnaltrexone (MNTX)
  Interventions: Drug: methylnaltrexone

INTERVENTIONS:
Drug: methylnaltrexone

SUMMARY:
This open-label study assesses the single-dose pharmacokinetics of intravenously-administered MNTX in healthy adult male and female subjects in the absence of, and in the presence of, orally-administered cimetidine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between the ages of 18 and 45
2. Subjects who are non-smokers
3. Subjects with body weights with range of 154-220 lbs.

Exclusion Criteria:

1. Females who are pregnant or lactating
2. Subjects with a history of any clinically significant disease or condition affecting a major organ system
3. Subjects with ECG abnormalities
4. Subjects who have tested positive for hepatitis B, hepatitis C or HIV
5. Subjects who have had a diagnosis of alcohol or substance dependence with the past 12 months
6. Subjects with positive urine results for drugs of abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of MNTX prior to and following multi-dose cimetidine regimen | 7 days
  To assess the potential effects of cimetidine on the pharmacokinetics of MNTX

SECONDARY OUTCOMES:
Area under the plasma concentration (AUC) of MNTX prior to and following a multi-dose cimetidine regimen | 7 days
  To assess the potential effects of cimetidine on the pharmacokinetics of MNTX
Half-life of MNTX prior to and following a multi-dose cimetidine regimen | 7 days
  To assess the potential effects of cimetidine on the pharmacokinetics of MNTX
Clearance (both total and renal)of MNTX prior to and following a multi-dose cimetidine regimen | 7 days
  To assess the potential effects of cimetidine on the pharmacokinetics of MNTX
Volume of distribution of MNTX prior to and following a multi-dose cimetidine regimen | 7 days
  To assess the potential effects of cimetidine on the pharmacokinetics of MNTX
Number of subject with adverse events as measured before, during, and after administration of cimetidine | 7 days
  To assess the potential effects of cimetidine on safety, and tolerability of MNTX

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States